CLINICAL TRIAL: NCT06621693
Title: Effect of Neuromuscular Electrical Stimulation on Phrenic Nerve Regeneration Post Cardiac Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Atef Abd El Fatah, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005299
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Post-cardiac Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical diaphragmatic stimulation intervention and traditional physiotherapy group (Experimental): This group will receive transcutaneous electrical diaphragmatic stimulation intervention and traditional physiotherapy three times per week for 4 weeks
  Interventions: Device: Transcutaneous electrical diaphragmatic stimulation intervention; Other: traditional physiotherapy program
- Traditional physiotherapy group (Active Comparator): This group will receive traditional physiotherapy only, three times per week for 4 weeks
  Interventions: Other: traditional physiotherapy program

INTERVENTIONS:
Device: Transcutaneous electrical diaphragmatic stimulation intervention — It will be applied on diaphragm, 30 min per session ,3 days/week for 4 weeks at a stimulation frequency of 30 Hz, pulse width of 400 μs, the intensity was gradually increased until visible muscle contraction was observed.
  Arms: Transcutaneous electrical diaphragmatic stimulation intervention and traditional physiotherapy group
Other: traditional physiotherapy program — The participants will receive traditional physiotherapy ( postural drainage, percussion , diaphragmatic breathing, phase 1 cardiac Rehabilitation and balance training ) three times per week for 4 weeks

SUMMARY:
This study will be conducted to investigate the effect of neuromuscular electrical stimulation on phrenic regeneration post cardiac surgery

DETAILED DESCRIPTION:
Phrenic nerve injury post cardiac surgery is a serious problem closely related to frequent respiratory complications. It has been associated with diaphragm dysfunction, pneumonia and difficulty weaning from mechanical ventilation in critical ill patients.

Neuromuscular electrical stimulation (NMES) is commonly used in physical therapy to increase muscle strength and promote muscle hypertrophy.

There is increased flow of patients after heart surgery in kasr Aini hospital who suffers from respiratory complication due to phrenic nerve injury so the hospitalization period of them increased which make economic burden in health insurance services with decreased level of quality of life that is the most concern as to improve patient status and relief this burden. So this study aims to decrease respiratory complication and improve phrenic nerve regeneration by using neuromuscular electrical stimulation as a safe, noninvasive , inexpensive and virtually risk free method.

ELIGIBILITY:
Inclusion Criteria:

* Patients post cardiac surgery (coronary artery bypass graft, valve repair or replacement ).
* Patients referred by physician.
* Medically stable patients.
* Both genders
* Ages from 25 to 45
* BMI 25-29.9 kg/m2
* Able to understand the requirements of the study.
* Conscious patient and respond to verbal commands.

Exclusion Criteria:

Participants will be excluded if they meet one of the following criteria:

* Patients with rib fracture.
* Patients developing lung cancer.
* Patients have dementia.
* Patients on mechanical ventilator after 24 hours
* Metabolically unstable chronic illness

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-04 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Phrenic nerve conduction study: motor latency | 4 weeks
  Nihon Kohden Neuropak M1 MEB-9200 EMG machine, made in Japan will be used to measure phrenic nerve conduction study.
  Motor latency is the impulse traveled from the stimulation site to the recording site is called latency and it is measured in milliseconds (ms). its normal value: (5.74ms -7.10 ms).
Phrenic nerve conduction study: Amplitude | 4 weeks
  Nihon Kohden Neuropak M1 MEB-9200 EMG machine, made in Japan will be used to measure phrenic nerve conduction study.
  Amplitude represents the maximal action potential depolarization and voltage gradient for all depolarized fibers of the phrenic nerve. it is measured in microvolt or millivolt (mv). its normal value: (0.47 mv-0.83 mv).

CONTACTS AND LOCATIONS:
Overall Officials: Hala R. Mahmoud, professor, Study Director — Cairo University; Nagwa M. Badr, professor, Study Chair — Cairo University
Locations (1):
- Hala Atef Abdel Fattah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol